CLINICAL TRIAL: NCT01111630
Title: Compare the Hemoglobin and Hematocrit Variability Between Once & Three Times Weekly Erythropoietin Therapy for the Anemia in Patients With Maintenance Dialysis
Brief Title: Study of Erythropoietin (EPO) Administration Schedule
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CWP_RCM_R01
Record Dates: First submitted 2010-04-25; First posted 2010-04-27 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Renal Failure; Anaemia
Keywords: chronic renal failure; Anaemia
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- once weekly (Experimental)
  Interventions: Drug: recomon (Epoetin Beta)
- three times weekly (Active Comparator)
  Interventions: Drug: recomon (Epoetin Beta)

INTERVENTIONS:
Drug: recomon (Epoetin Beta) — administer once weekly
  Arms: once weekly
Drug: recomon (Epoetin Beta) — administer three times weekly
  Arms: three times weekly

SUMMARY:
The purpose of this study is to compare the hemoglobin and hematocrit variability between once and three times weekly erythropoietin therapy for the anemia in patients with maintenance dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80.
* Dialysis for at least 3 months.
* Epoetin treatment for the last 3 months.
* Baseline hemoglobin (Hb) value of >= 9.0 g/dL and < 13.0 g/dL.
* Baseline mean weekly epoetin maintenance dose ≤ 12,000 IU
* Patients who agree to participate in this study in writing.

Exclusion Criteria:

* Hemoglobinopathies, i.e. sickle cell disease, thalassemia of all types.
* Hemolysis as defined
* Gastrointestinal bleeding necessitating treatment (medication, transfusion) within the last 3 months.
* Patients with uncontrolled hypertension.
* Acute infection of unstable systemic inflammatory disease.
* Current malignant disease.
* High likelihood of early withdrawal or interruption of the study (e.g. severe diseases within the last 3 months, such as myocardial infarction, unstable angina, stroke, deep venous thrombosis).
* Life expectancy below 12 months.
* Planned elective surgery during the study period.
* Blood transfusions within the last 3 months.
* Pregnancy and lactation.
* Other conditions regarded as unsuitability by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The hemoglobin variability between once & three times weekly administration | 24 weeks

SECONDARY OUTCOMES:
The hematocrit variability between once & three times weekly administration | 24 weeks
Mean value of Hb and Hct between once & three times weekly administration | 24 weeks
Drop out rate during dose fix period | 24 weeks
Mean value of Hb and Hct during dose fix period | 24 weeks
Variability of Hb and Hct during dose fix period | 24weeks
Weekly oetin-beta maintenance dose between once & three times weekly administration | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SugKyun Shin, Ph.D., Principal Investigator — National Health Insurance Service Ilsan Hospital
Locations (1):
- NHIC Ilsan Hospital, Seoul, South Korea